CLINICAL TRIAL: NCT02232906
Title: Pilot Open Label Study to Evaluate Intravenous Ferric Carboxymaltose (Ferinject ®) in Patients With CKD (Pre-dialysis) With Anemia Treated With Epo and Oral Iron in Buenos Aires, Argentina
Brief Title: Switch From Oral Iron to Intravenous Ferric Carboxymaltose in Non-dialysis Chronic Kidney Disease (CKD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Aleman (Other)
Collaborators: Vifor Pharma (Industry)
Responsible Party: Principal Investigator, Jorge Eduardo Toblli, Full Professor of Medicine at University of Buenos Aires, Argentina, and Director of the Laboratory of Experimental Medicine, Hospital Alemán, Buenos Aires., Hospital Aleman
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FCM-ND-CKD 2012
Record Dates: First submitted 2014-08-31; First posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-09

CONDITIONS: Iron Deficiency; Anaemia
Keywords: Chronic kidney disease; CKD; non-dialysis-dependent; ND-CKD; Erythropoiesis-stimulating agent; Ferric carboxymaltose; Iron
MeSH Terms: conditions — Iron Deficiencies; Anemia; Renal Insufficiency, Chronic | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- intravenous ferric carboxymaltose (Experimental)
  Interventions: Drug: intravenous ferric carboxymaltose

INTERVENTIONS:
Drug: intravenous ferric carboxymaltose — Ferric carboxymaltose (FCM) dose of 1,000 mg iron, followed by a 6-month ESA/FCM maintenance regimen (target: Hemoglobin 120 g/L, transferrin saturation >20%)
  Other Names: Ferinject, Injectafer

SUMMARY:
Investigation whether a switch from oral iron to intravenous ferric carboxymaltose can reduce dose requirements of erythropoiesis-stimulating agents (ESA) and improve Hb levels and iron status in adult patients with non-dialysis-dependent CKD who were on a stable ESA/oral iron schedule for 6 months prior to enrolment.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Creatinine clearance ≤40 mL/min
* Hemoglobin 110-120 g/L
* Serum ferritin <100 µg/L or transferrin saturation <20%
* Monthly treatment with ESA and oral iron for at least six months before enrolment

Exclusion Criteria:

* Other obvious cause of acute or chronic anemia than iron deficiency
* Expectation to require hemodialysis within the next six months
* Short life expectancy (<1 year)
* Pregnancy
* Decompensated heart failure
* History of allergic reactions to iron preparations and/or anaphylaxis from any cause
* Requirement of blood transfusions
* Chronic decompensated mental disorder or dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-03; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
ESA dose requirement during the observation period after the switch from oral iron to intravenous ferric carboxymaltose treatment | 6 months

SECONDARY OUTCOMES:
Anaemia and iron status | 6 months
  Hemoglobin, mean corpuscular volume, serum ferritin and transferrin saturation were assessed at baseline and monthly until end of study
Number of hospitalizations | 6 months
Number of transfusions | 6 months
Number of adverse reactions | 6 months
Creatinine clearance at baseline and then bi-monthly until end of study as marker of renal function | 6 months
Proteinuria at baseline and then bi-monthly until end of study as marker of renal function | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E Toblli, Prof., MD, Principal Investigator — Hospital Aleman
Locations (1):
- Hospital Alemán, Buenos Aires, Argentina

REFERENCES:
- [Derived] Toblli JE, Di Gennaro F. Switching patients with non-dialysis chronic kidney disease from oral iron to intravenous ferric carboxymaltose: effects on erythropoiesis-stimulating agent requirements, costs, hemoglobin and iron status. PLoS One. 2015 Apr 30;10(4):e0125528. doi: 10.1371/journal.pone.0125528. eCollection 2015. PMID 25928811